CLINICAL TRIAL: NCT05829954
Title: The Body Awareness and Its Relationship Musculoskeletal Problems in Dentistry Students and Dentists
Brief Title: Body Awareness in Dentistry Students and Working Dentists
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, HATİCE ÇETİN, Assist, Prof, Hacettepe University
Other Study IDs: DBA123
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Musculoskeletal Diseases; Body Image; Dentistry
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1st dentistry students: 1st dentistry students
  Interventions: Other: questionnaire
- Intern dentistry students: 5th dentistry students
  Interventions: Other: questionnaire
- working dentists: dentists who have worked for at least two years
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — All questionnaire were obtained via online survey system.

SUMMARY:
The current study aims to comparison the body awareness and musculoskeletal problems of 1st dentistry students, intern students and working dentists and also investigate the factors affecting the body awareness over the years in dentistry profession.

DETAILED DESCRIPTION:
Dentists also have the highest prevalence among the occupational groups providing health services. More than 60% of dentists have pain in at least one of their body parts.Pain due to musculoskeletal disorders can affect body awareness of person have chronic pain. Body awareness is known as the capacity to distinguish body parts and has an important role in promoting well-coordinated movements. The current study aims to comparison the body awareness and musculoskeletal problems of 1st dentistry students, intern students and working dentists and also investigate the factors affecting the body awareness over the years in dentistry profession.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are being between the ages of 18 and 65 and had been practising dentistry for more than two years for dentists group.

Exclusion Criteria:

* The exclusion criteria are had a surgical history of vertebral column or any neurological or inflammatory disorders or trauma history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dentistry students and dentists
Sampling Method: Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnaire | At baseline
  The questionnaire includes physical, emotional and social elements about the sensitivity of a person to normal or abnormal body conditions and processes and questioning the sensitivity to physical reactions. Participants were asked to rate between 1 and 7 for each of the 18 statements (1=Not at all relevant to me, 7=Very appropriate to me). The total score ranges from 18 to 126. As the score increases, BA increases.
Nordic Musculoskeletal Questionnaire | At baseline
  The questionnaire, was developed by Nordic Council of Ministers in 1987, evaluates musculoskeletal pain intensities of nine body parts; neck, shoulder, elbow, wrist, upper and lower back, hip, knee and ankle in the last seven days. Pain intensities were questioned according to Visual Analog Scale.

SECONDARY OUTCOMES:
Oswestry Disability Index | At baseline
  Oswestry Disability Index assesses ten different aspects of disability (pain, personal care, lifting, sitting, standing, sleeping, sex life, social life, walking, and travelling). Each parameter is scored from 0 to 5 (0; no functional limitation due to pain, 5; a significant functional disability due to low back pain). This questionnaire is scored using a global percentage score. The obtainable maximum score is 50.
Neck Disability Index | At baseline
  It is the most commonly used outcome measure for neck pain and it contains 10 subsections consisting of severity of pain, personal care, lifting, reading, headache, concentration, work, driving, sleeping, and leisure activities. The questions are measured between 0-5 points (0: no pain and functional limitation, 5: worst pain and maximal limitation). The numeric response for each item is summed for a score varying from 0 to 100.
Hospital Anxiety-Depression Scale | At baseline
  The Hospital Anxiety and Depression Scale is used for assessing the anxiety and depression levels of the patients. The items were scored from 0-3 (0: not present, 3: considerable). The cutoff scores were 10 for anxiety and 7 for depression. A high score indicates the risk of anxiety and depression.
Tampa Scale of Kinesiophobia | At baseline
  Tampa Kinesiophobia Scale was used for evaluating kinesiophobia. Each item was scored on a Likert scale (1; Strongly disagree, 4; Totally agree) was used. Scores between 17 and 68 are obtained from the questionnaire. The higher score indicated a higher kinesiophobia.
Nottingham Health Profile: | At baseline
  It contains scales for physical mobility, social isolation, sleep, pain, emotional reactions and energy. The total score changes between 0-100 for each scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Bilgin, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No